CLINICAL TRIAL: NCT04382690
Title: Surveys of the Behavioral Determinants That May Influence People's Hand-hygiene and Environment Disinfecting in Different Countries
Brief Title: Behavioral Determinants That May Influence People's Hand-hygiene and Environment Disinfecting
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Responsible Party: Principal Investigator, Kelly Ann Schmidtke, Assistant Professor, University of Warwick
Other Study IDs: 8304
Record Dates: First submitted 2020-04-25; First posted 2020-05-11 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Hygiene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- India: People residing in India
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions
- United Kingdom: People residing in the United Kingdom
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions
- China: People residing in China
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions
- Australia: People residing in Australia
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions
- South Africa: People residing in South Africa
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions
- Indonesia: People residing in Indonesia
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions
- Saudi Arabia: People residing in Saudi Arabia
  Interventions: Behavioral: All participants will be asked to respond to the same survey questions

INTERVENTIONS:
Behavioral: All participants will be asked to respond to the same survey questions — All participants will be asked to respond to the same survey questions

SUMMARY:
An anonymous online survey will be conducted to measure the barriers and facilitators parents and teachers experience to positively influencing children's hand-hygiene. A sub-section of the survey will also examine the barriers and facilitators they experience to surface cleaning. The final survey will be conducted with participants from Australia, China, India, Indonesia, Saudi Arabia, South Africa, and the United Kingdom. The data collected will be completely anonymous and there are no sensitive questions. The primary and secondary analyses will focus on the hand-hygiene items to examine the survey's internal and external validity. The results will inform a future school-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older;
* identify as a female or male; and
* be either a teacher or parent of children between 5 and 10 years old.

Exclusion Criteria:

* be 17 years or younger;
* not identify as a female or male; and
* not be a teacher or parent of children between 5 and 10 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be residents of one of the following countries: Australia, China, India, Indonesia, Saudi Arabia, South Africa, and the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 3975 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Theoretical Domains Framework Barriers/Facilitators | Reported during the survey on Day 1
  Participants' agreements with survey statements about the barriers and facilitators they expereince to positively influecing children's hand hygeine and surface cleaning. Each response is given on a 5 point scale from strongly disagree to strongly agree. Some statements will be reverse scored.

SECONDARY OUTCOMES:
Self-reported confience in positively influencing children's hygeine when they are watching | Reported during the survey on Day 1
  Participants' responses to the following question: When your [children/pupils] can see you watching them, what percentage of the time do they wash their hands with soap and water after going to the toilet and before eating? [response options 0% - 100%]
Self-reported confience in positively influencing children's hygeine when they are not watching | Reported during the survey on Day 1
  Participants' responses to the following question: When your [children/pupils] cannot see you watching them, what percentage of the time do they wash their hands with soap and water after going to the toilet and before eating?'[response options 0 - 100%]
Self-reported hygiene | Reported during the survey on Day 1
  Participants' responses to the following question: What percentage of the time do you wash your own hands with soap and water after going to the toilet and before eating? [response options 0-100%]

OTHER OUTCOMES:
Country | Reported during the survey on Day 1
  The country participants live in, either: India, the United Kingdom, China, Australia, South Africa, Indonesia, or Saudi Arabia
Gender | Reported during the survey on Day 1
  What gender participants identify with: Male, Female, Other/prefer not to say
Age | Reported during the survey on Day 1
  Participants' ages: 18 - 30 years old, 31 - 40 years old, 40 - 50 years old, 50 - 60 years old, 61 - 70 years old, or 70 or more years old
Parent or Teacher | Reported during the survey on Day 1
  Participants' life roles that might help them influence children's hygiene: Mum, Dad, Teacher
Occupation | Reported during the survey on Day 1
  Participants' employment status: Work full-time, Work part-time, Retired, Full-time, Home-maker / parent, Student, Unemployed, or Other

CONTACTS AND LOCATIONS:
Locations (1):
- University of Warwick, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT04382690/Prot_SAP_ICF_000.pdf